CLINICAL TRIAL: NCT05089474
Title: A First in Human Clinical Trial to Evaluate the Safety and Effectiveness of the STREAMLINE SURGICAL SYSTEM in Patients With Open-Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New World Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DF6-CL-20-01
Record Dates: First submitted 2021-10-13; First posted 2021-10-22 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-01

CONDITIONS: Open Angle Glaucoma
Keywords: Open Angle Glaucoma, IOP, viscoelastic
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Streamline (Experimental): Streamline Surgical System
  Interventions: Device: Streamline Surgical System

INTERVENTIONS:
Device: Streamline Surgical System — The Streamline System is a device that delivers viscoelastic into Schlemm's Canal.

SUMMARY:
A prospective, nonrandomized, open label study to evaluate the safety and IOP lowering effectiveness of the Streamline Surgical System, in patients with mild-to-moderate open angle glaucoma undergoing cataract surgery.

DETAILED DESCRIPTION:
A prospective, nonrandomized, open label study to evaluate the safety and IOP lowering effectiveness of the Streamline Surgical System, a viscoelastic delivery device, in patients with mild-to-moderate open angle glaucoma undergoing cataract surgery. This is a 12 month study conducted outside the US. Approximately 60 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and execute written informed consent
2. Males or female subjects at least 22 years of age.
3. Subjects qualifying for cataract surgery
4. Subjects diagnosed with mild to moderate open-angle glaucoma in at least one eye currently treated with 1-3 topical IOP-lowering medications
5. Subjects with diagnosis of open-angle glaucoma in at least one eye with an unmedicated IOP of 21-36 mmHg

Exclusion Criteria:

1. Women of child-bearing potential
2. Modified Shaffer angle grade < 2
3. Patients with severe or advanced glaucoma
4. Intraocular surgery within the last 6 months or laser surgery within the last 3 months
5. BCVA worse than 20/80 in either eye
6. Patients with a previous peripheral iridotomy.
7. Ocular infection or inflammation within the last 6 months.
8. Any medication that would be contraindicated for a glaucoma surgical procedure.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
proportion of unmedicated eyes with IOP reduction of > 20% from Baseline at Month 12. | 12 months
  Primary Endpoint

SECONDARY OUTCOMES:
Adverse Events | 12 months
  Assess intraoperative and post operative AEs
Mean IOP change | 12 months
  Mean IOP change in unmedicated IOP from baseline to M12
Number of topical glaucoma medications | 12 months
  Number of topical glaucoma medications used at screening compared to Month 12

CONTACTS AND LOCATIONS:
Locations (3):
- Clinica 20/20, San José, CR, Costa Rica
- Centro Laser, Santo Domingo, DR, Dominican Republic
- Clinica Laser y Ultrasonido Ocular de Puebla, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No